CLINICAL TRIAL: NCT01453127
Title: DaTSCAN Imaging in Aging and Neurodegenerative Disease
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley Boeve, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-001999
Record Dates: First submitted 2011-09-28; First posted 2011-10-17 (Estimated); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Dementia; Parkinsonism; Mild Cognitive Impairment; REM Sleep Behavior Disorder
Keywords: dementia; parkinsonism; mild cognitive impairment; REM sleep behavior disorder
MeSH Terms: conditions — Dementia; Parkinsonian Disorders; Cognitive Dysfunction; REM Sleep Behavior Disorder | interventions — ioflupane; Tomography, Emission-Computed, Single-Photon; Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (8):
- Alzheimer's Disease (Experimental): Alzheimer's Disease
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Dementia with Lewy Bodies (Experimental): Dementia with Lewy Bodies
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Frontotemporal Dementia (Experimental): Frontotemporal Dementia
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Parkinson's Disease (Experimental): Parkinson's Disease
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Corticobasal Degeneration (Experimental): Corticobasal Degeneration
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Essential Tremor (Experimental): Essential Tremor
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- Mild Cognitive Impairment (Experimental): Mild Cognitive Impairment
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan
- REM sleep behavior disorder (Experimental): REM sleep behavior disorder
  Interventions: Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan); Device: Single photon emission computed tomography (SPECT) scan

INTERVENTIONS:
Drug: I-123 Ioflupane solution injection prior to SPECT scan (DaTscan) — I-123 Ioflupane solution for injection into a living test subject. The iodine introduced during manufacture is a radioactive isotope, I-123, and it is the properties of this isotope that makes the solution visible to a gamma camera on SPECT imaging. I-123 has a half-life of approximately 13 hours and a gamma photon energy of 159 keV making it an good radionuclide for medical imaging. DaTscan is administered by intravenous cannula. The scan is carried out 3-6 hours post injection.
Device: Single photon emission computed tomography (SPECT) scan — Single-photon emission computed tomography(SPECT)is a nuclear medicine tomographic imaging technique using gamma rays. It is very similar to conventional nuclear medicine planar imaging using a gamma camera. However, it is able to provide true 3D information. This information is typically presented as cross-sectional slices through the patient, but can be freely reformatted or manipulated as required.

SUMMARY:
The investigators propose using DaTscan in patients with REM sleep behavior disorder (RBD), mild cognitive impairment (MCI), Parkinson's disease (PD), dementia with Lewy bodies (DLB), Alzheimer's disease (AD), and other neurodegenerative syndromes and disorders, to test several hypotheses - some confirmatory, and some novel. Such use will provide new data on the potential clinical and research utility of DaTscan in neurodegenerative diseases. The findings on DaTscan will be correlated with clinical diagnoses and other multimodal imaging studies (e.g., MRI, MRS, FDG-PET, and amyloid-PET) to enhance our understanding of neurodegenerative diseases.

DETAILED DESCRIPTION:
Lewy body disease (LBD) is one of the most common neurodegenerative diseases and second only to Alzheimer's disease in terms of prevalence, disability, and societal/financial burden. The phenotypic variability of LBD is striking, as it can manifest as the well-known disorder of Parkinson's disease without (PD) and with dementia (PDD), as well as DLB, MCI, REM sleep behavior disorder (RBD), pure autonomic failure (PAF), and other syndromes.

One biomarker which is both highly sensitive and specific for evolving LBD in the setting of dementia is DaTscan [Ioflupane (123I)] imaging, in which loss of functional dopaminergic neuron terminals in the striatum as assessed by DaTscan reflects underlying LBD in those with dementia and particularly dementia with Lewy bodies (DLB). DaTscan is the one of the first radiopharmaceutical agents available to detect DaT distribution within the brain. DaTscan imaging involves injection of the Ioflupane radioligand followed by imaging using a standard single photon emission computed tomography (SPECT) scanner. DaTscan provides visualization of the dopamine transporter (DaT) distribution within the striata (i.e., striatal uptake, or striatal signal) by SPECT imaging in patients presenting with symptoms or signs suggestive of dopaminergic neurodegeneration.

Most DaTscan studies published to date have been conducted in centers outside of the US. DaTscan has not been studied in the syndrome of MCI, and minimally in corticobasal degeneration (CBD). Very little normative data exists in the aged population either.

The FDA-approved indication is to assist in the evaluation of adult patients with suspected Parkinsonian syndromes (PS). In these patients, DaTscan may be used to help differentiate essential tremor from tremor due to Parkinsonian syndromes (such as idiopathic Parkinson's disease, multiple system atrophy and progressive supranuclear palsy). DaTscan will be used as an adjunct to other diagnostic evaluations. Identifying dopaminergic dysfunction is also important in other settings such as those with cognitive impairment with or without parkinsonism, and in subjects with REM sleep behavior disorder. The findings on DaTscan in subjects with these various disorders will be correlated with clinical diagnoses and other multimodal imaging studies (e.g., MRI, MRS, FDG-PET, and amyloid-PET) to enhance our understanding of neurodegenerative diseases. A subset of subjects will undergo a 2nd DaTscan at least 1 year after the initial scan was performed to determine if changes over time provide any prognostic information.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the syndromes of interest using established criteria
* Age 40-90 inclusive
* MMSE score above 10
* No active medical disorder that could preclude participation
* Stable medication regimen over previous four weeks
* Absence of certain medications that could significantly impact the DaTscan findings
* For those with dementia, caregiver that is with the patient at least 4 hours/day for at least 5 days per week
* For those with dementia, or severe parkinsonism, patient and caregiver willing and able to participate in all study-related procedures
* Patient is capable of giving informed consent, or if appropriate, has caregiver capable of giving consent on the subject's behalf.

Exclusion Criteria:

* Does not fulfill criteria for any of the desired diagnoses
* Age <40 or >90
* Women with intact uterus and not post-menopausal unless pregnancy test performed at screening is negative
* Women who are pregnant or are breast-feeding an infant
* MMSE score <10
* Active medical disorder that could preclude participation in this protocol

  * Hypersensitivity to the radioligand, cocaine, or iodine (including seafood allergy)
  * Myocardial infarction or cerebral infarct over preceding year, stable or unstable angina, known symptomatic coronary artery disease
  * Renal or liver disease viewed by the physician to be too severe to warrant DaTscan infusion/imaging
  * History of significant alcohol or drug abuse
  * Any other medical disorder considered by the study physicians as inappropriate for this protocol
* Patient or caregiver unwilling or unable to participate in all study-related procedures
* Caregiver is not with a patient with dementia or severe parkinsonism at least 4 hours/day for at least 5 days/week
* Patient or caregiver unwilling or unable to provide informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlate the DaTscan findings with clinical diagnosis | Participants will be followed to 1-3 days after scan.
  The primary endpoint is to correlate the DaTscan findings with clinical diagnosis

SECONDARY OUTCOMES:
Safety of DaTscan imaging | Participants will be followed for 1-3 days after scan.
  The primary safety/tolerability endpoint relates to side effects associated with DaTscan imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Boeve, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Arnaldi D, Mattioli P, Raffa S, Pardini M, Massa F, Iranzo A, Perissinotti A, Ninerola-Baizan A, Gaig C, Serradell M, Munoz-Lopetegi A, Maya G, Liguori C, Fernandes M, Placidi F, Chiaravalloti A, Sonka K, Dusek P, Zogala D, Trnka J, Boeve BF, Miyagawa T, Lowe VJ, Miyamoto T, Miyamoto M, Puligheddu M, Figorilli M, Serra A, Hu MT, Klein JC, Bes F, Kunz D, Cochen De Cock V, de Verbizier D, Plazzi G, Antelmi E, Terzaghi M, Bossert I, Kulcsarova K, Martino A, Giuliani A, Pagani M, Nobili F, Morbelli S; International REM Sleep Behavior Disorder Study Group. Presynaptic Dopaminergic Imaging Characterizes Patients with REM Sleep Behavior Disorder Due to Synucleinopathy. Ann Neurol. 2024 Jun;95(6):1178-1192. doi: 10.1002/ana.26902. Epub 2024 Mar 11. PMID 38466158
- [Result] Jung Y, Jordan LG 3rd, Lowe VJ, Kantarci K, Parisi JE, Dickson DW, Murray ME, Reichard RR, Ferman TJ, Jones DT, Graff-Radford J, Savica R, Machulda MM, Fields JA, Allen LA, Drubach DA, St Louis EK, Silber MH, Jack CR Jr, Knopman DS, Petersen RC, Boeve BF. Clinicopathological and 123I-FP-CIT SPECT correlations in patients with dementia. Ann Clin Transl Neurol. 2018 Jan 24;5(3):376-381. doi: 10.1002/acn3.521. eCollection 2018 Mar. PMID 29560382
- [Result] Chen Q, Lowe VJ, Boeve BF, Przybelski SA, Miyagawa T, Senjem ML, Jack CR Jr, Lesnick TG, Kremers WK, Fields JA, Min HK, Schwarz CG, Gunter JL, Graff-Radford J, Savica R, Knopman DS, Jones D, Ferman TJ, Graff-Radford NR, Petersen RC, Kantarci K. beta-Amyloid PET and 123I-FP-CIT SPECT in Mild Cognitive Impairment at Risk for Lewy Body Dementia. Neurology. 2021 Feb 22;96(8):e1180-e1189. doi: 10.1212/WNL.0000000000011454. PMID 33408148
- [Result] Maltais DD, Jordan LG, Min HK, Miyagawa T, Przybelski SA, Lesnick TG, Reichard RR, Dickson DW, Murray ME, Kantarci K, Boeve BF, Lowe VJ. Confirmation of 123I-FP-CIT SPECT Quantification Methods in Dementia with Lewy Bodies and Other Neurodegenerative Disorders. J Nucl Med. 2020 Nov;61(11):1628-1635. doi: 10.2967/jnumed.119.239418. Epub 2020 Mar 20. PMID 32198310
- [Result] Miyagawa T, Przybelski SA, Maltais D, Min HK, Jordan L, Lesnick TG, Chen Q, Graff-Radford J, Jones D, Savica R, Knopman D, Petersen R, Kremers WK, Forsberg LK, Fields JA, Ferman TJ, Allen L, Parisi J, Reichard RR, Murray M, Dickson D, Boeve BF, Kantarci K, Lowe VJ. The value of multimodal imaging with 123I-FP-CIT SPECT in differential diagnosis of dementia with Lewy bodies and Alzheimer's disease dementia. Neurobiol Aging. 2021 Mar;99:11-18. doi: 10.1016/j.neurobiolaging.2020.12.009. Epub 2020 Dec 15. PMID 33422890
- [Result] Arnaldi D, Chincarini A, Hu MT, Sonka K, Boeve B, Miyamoto T, Puligheddu M, De Cock VC, Terzaghi M, Plazzi G, Tachibana N, Morbelli S, Rolinski M, Dusek P, Lowe V, Miyamoto M, Figorilli M, Verbizier D, Bossert I, Antelmi E, Meli R, Barber TR, Trnka J, Miyagawa T, Serra A, Pizza F, Bauckneht M, Bradley KM, Zogala D, McGowan DR, Jordan L, Manni R, Nobili F. Dopaminergic imaging and clinical predictors for phenoconversion of REM sleep behaviour disorder. Brain. 2021 Feb 12;144(1):278-287. doi: 10.1093/brain/awaa365. PMID 33348363
- [Result] Diaz-Galvan P, Miyagawa T, Przybelski SA, Lesnick TG, Senjem ML, Jack CR Jr, Forsberg LK, Min HK, St Louis EK, Savica R, Fields JA, Benarroch EE, Lowe V, Petersen RC, Boeve BF, Kantarci K. Brain glucose metabolism and nigrostriatal degeneration in isolated rapid eye movement sleep behaviour disorder. Brain Commun. 2023 Feb 2;5(1):fcad021. doi: 10.1093/braincomms/fcad021. eCollection 2023. PMID 36844148
- See also: Mayo Clinic Clinical Trials - Lewy Body Disease — https://www.mayo.edu/research/clinical-trials/search-results?keyword=lewy&studySiteStatusesGrouped=Open/Status%20Unknown